CLINICAL TRIAL: NCT05338151
Title: Promoting Alcohol Treatment Engagement Post-hospitalization With Brief Intervention, Medications and CBT4CBT: A Randomized Clinical Trial in a Diverse Patient Population.
Brief Title: Promoting Alcohol Treatment Engagement Post-hospitalization
Acronym: ENHANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000031874; 1R01AA029820-01 (NIH)
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
Keywords: CBT4CBT; Brief Negotiated Interview (BNI); Medication for alcohol use disorder (MAUD); Phosphatidylethanol (PEth)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief Negotiated Interview (with referral and telephone booster) alone (Other): All participants will receive BNI with referral and a 15-20 minute telephone booster delivered by a trained Health Promotion Advocate (HPA) at 2 weeks. The purpose of the BNI is to assist patients in recognizing and changing levels of alcohol consumption that pose health risks. The main goals of the BNI are to: 1) lessen ambivalence about reducing alcohol use; and 2) negotiate strategies for change. During BNI, the HPA will: 1) Raise the subject of alcohol; 2) Provide feedback: review the patient's alcohol consumption, make a connection to the patient's medical condition and reason for hospitalization; review guidelines for lower risk alcohol use; 3) Enhance motivation: have the patient identify on a readiness change ruler and develop discrepancy; and 4) Negotiate and Advise: negotiate goal, give advice, have patient complete drinking agreement; summarize and arrange follow-up.
  Interventions: Behavioral: Brief Negotiated Interview (BNI)
- BNI+MAUD (Active Comparator): For either BNI+facilitated provision of MAUD or BNI+facilitated provision of MAUD+CBT4CBT, the HPA will provide education and counseling regarding MAUD as part of the BNI to the participant and communicate to the primary medical team that MAUD is indicated. The specific MAUD chosen will be made at the discretion of the patient and the primary medical team with recommendations from the study physicians, with a goal of prioritizing FDA approved medications. Participants will be encouraged to initiate (or receive as in the case of injectable naltrexone) MAUD prior to discharge and will be provided a prescription for a 30-day supply. Medications will be obtained through regular means and not provided directly through the study. During the BNI telephone booster, the HPA will inquire about and address any barriers to MAUD and encourage continued adherence.
  Interventions: Behavioral: BNI+facilitated provision of MAUD
- BNI+MAUD+CBT4CBT (Experimental): Participants randomized to BNI+facilitated provision of MAUD+CBT4CBT will be given a username and password to access the web-based program and be encouraged to begin accessing the program during their hospitalization. The HPA will assist each participant with login during the first session and be available to answer any questions. Participants will be asked to complete no more than two modules per week, with an expectation of completing all seven modules by the end of the 34-day post-discharge. The program tracks, for each participant, time logged onto the program, modules accessed, progress through the program from session to session, completion of homework assignments, and learning of CBT principles through brief quizzes. Participants will be allowed to repeat modules as desired. During the BNI telephone booster, the HPA will inquire about engagement with CBT4CBT, address any questions and problems with the program, and encourage practice of coping activities (i.e., homework).
  Interventions: Behavioral: Brief Negotiated Interview BNI+facilitated provision of MAUD+CBT4CBT

INTERVENTIONS:
Behavioral: Brief Negotiated Interview (BNI) — Brief Negotiated Interview (with referral and telephone booster) alone
  Arms: Brief Negotiated Interview (with referral and telephone booster) alone
Behavioral: BNI+facilitated provision of MAUD — Brief Negotiated Interview (BNI)+ Medication for Alcohol Use Disorder (MAUD)
  Arms: BNI+MAUD
Behavioral: Brief Negotiated Interview BNI+facilitated provision of MAUD+CBT4CBT — Brief Negotiated Interview (BNI)+Medication for Alcohol Use Disorder (MAUD)+Computer Based Treatment for Cognitive Behavioral Treatment (CBT4CBT)
  Arms: BNI+MAUD+CBT4CBT

SUMMARY:
This study is a 3-arm randomized clinical trial to evaluate the effectiveness of hospital-initiated Alcohol Use Disorder treatment, involving a Brief Negotiated Interview (with referral and telephone booster) alone, BNI+facilitated provision of MAUD, BNI+facilitated provision of MAUD+CBT4CBT on AUD treatment engagement, alcohol use and healthcare utilization.

DETAILED DESCRIPTION:
The proposed 3-arm randomized clinical trial will initiate interventions during hospitalization and evaluate outcomes at 34- and 90-days following hospital discharge to compare the effectiveness of 1) BNI, 2) BNI+facilitated provision of MAUD, and 3) BNI+facilitated provision of MAUD+CBT4CBT on AUD treatment engagement, alcohol consumption, and healthcare utilization among 450 racially and ethnically diverse hospitalized individuals with AUD.

Using a hybrid type 1 effectiveness-implementation design the investigators will also conduct an implementation- focused process evaluation to yield relevant data to inform future implementation, including process measures, clinician and staff (n=150) perspectives and cost effectiveness.

This proposed study is directly informed by rigorous prior research by this group and others demonstrating: 1) a need for new strategies to engage patients, particularly Black and Hispanic individuals, with AUD in treatment; 2) benefits of engaging patients in addiction treatment during acute care;3) benefits of MAUD and the potential to integrate its provision in general medical settings; and 4) benefits of CBT as an adjunct to MAUD with strong support for CBT4CBT across diverse populations

ELIGIBILITY:
Inclusion Criteria:

* hospitalized at Yale New Haven Hospital (YNHH)
* meet Diagnostic and Statistical Manual (DSM-5) criteria for a moderate to severe AUD (regardless of primary reason for hospitalization) consistent with clinical guidelines for MAUD initiation
* >1 heavy drinking day by TLFB in 30 days prior to hospitalization
* willing to consider MAUD
* willing and able to be contacted for follow-up
* provide written informed consent

Exclusion Criteria:

* have been engaged in formal AUD treatment in the past 30 days (i.e., excluding mutual help groups, such as Alcoholics Anonymous)
* meet DSM-5 criteria for untreated moderate to severe opioid use disorder
* self-reported or urine testing confirming pregnancy, nursing, or trying to conceive
* life-threatening or unstable medical, surgical, or psychiatric condition that prohibits study participation
* inability to provide >1 collateral contact for a friend or family member
* anticipate being unable to return for follow-up assessments for any reason, such as travel, incarceration, planned procedure
* inability to understand English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the percentage of participants engaged in AUD Treatment at the 34-day post hospital discharge timepoint, defined as any self-reported AUD treatment service assessed on the AUD Treatment Assessment. | Day 34 post hospital diacharge
  AUD Treatment Engagement Assessment is a self-report used to assess if participants have participated in different types of treatment engagement for alcohol use over 34 days. That data is verified by an outside source.

SECONDARY OUTCOMES:
Change from baseline in alcohol use by percentage of heavy drinking days at day 34 and 90. | Baseline, day 34 and day 90
  Change in alcohol use by percentage of heavy drinking days operationalized by the Timeline Followback (TLFB) method. TLFB is administered by an interviewer and involves asking clients to retrospectively estimate their alcohol and drug use 34 and 90 days prior to the interview date.
Change from baseline in alcohol use at days 34 and 90 using a Phosphatidylethanol (PEth) test | Baseline, day 34 and day 90
  Change from baseline in alcohol use at 34 and 90 days post discharge measured by PEth in the blood. PEth is a finger stick blood draw to detect alcohol use by detecting direct alcohol biomarkers in the bloodstream. A positive test indicates alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: E. Jennifer Edelman, MD, Principal Investigator — Yale University; Brian Kiluk, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Edelman EJ, Frankforter T, Rojas-Perez OF, Ablondi K, Castro C, Corvino J, Garcia I, Gordon DM, Jaramillo Y, Johnson NL, Jordan A, Nich C, Paris M Jr, Pagano D, Weimer MB, Williams EC, Kiluk BD. Promoting Race and Ethnic Diversity in a Hospital-Based Randomized Clinical Trial to Address Untreated Alcohol Use Disorder: Initial Lessons Learned. J Addict Med. 2025 May-Jun 01;19(3):334-337. doi: 10.1097/ADM.0000000000001400. Epub 2024 Nov 8. PMID 39514895
- [Derived] Edelman EJ, Rojas-Perez OF, Nich C, Corvino J, Frankforter T, Gordon D, Jordan A, Paris M Jr, Weimer MB, Yates BT, Williams EC, Kiluk BD. Promoting alcohol treatment engagement post-hospitalization with brief intervention, medications and CBT4CBT: protocol for a randomized clinical trial in a diverse patient population. Addict Sci Clin Pract. 2023 Sep 19;18(1):55. doi: 10.1186/s13722-023-00407-9. PMID 37726823